CLINICAL TRIAL: NCT04935164
Title: Comparative Study of Gender Dysphoria Phenomenology and Neurophysiology: Clinical and Experimental Exploration of Gender Identity Disorder
Brief Title: Comparative Study of Gender Identity Disorder Versus Control
Acronym: TRANSIDENT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03407-32
Record Dates: First submitted 2021-02-26; First posted 2021-06-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Gender Dysphoria, Adult
MeSH Terms: conditions — Gender Dysphoria | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Male patients with gender dysphoria: * male patients with gender dysphoria according to DSM-V criteria (axis I), confirmed by MINI evaluation
  * patients without psychotropic treatments
  * patients who do not benefit of hormone therapy
  * patients who have not yet received gender reassignment surgery
  * patients aged 18 to 60 years
  * patients with normal or corrected vision
  * patients without mental defect
  * patients without neurological impairment
  Interventions: Other: Psychiatric evaluations
- Female patients with gender dysphoria: * female patients with gender dysphoria according to DSM-V criteria (axis I), confirmed by MINI evaluation
  * patients without psychotropic treatments
  * patients who do not benefit of hormone therapy
  * patients who have not yet received gender reassignment surgery
  * patients aged 18 to 60 years
  * patients with normal or corrected vision
  * patients without mental defect
  * patients without neurological impairment
  Interventions: Other: Psychiatric evaluations
- Male volunteers without gender dysphoria: * male volunteer without gender dysphoria according to DSM-V criteria (axis I), confirmed by MINI evaluation
  * volunteer aged 18 to 60 years
  * volunteer with normal or corrected vision
  * volunteer without mental defect
  * volunteer without neurological impairment
  Interventions: Other: Psychiatric evaluations
- Female volunteers without gender dysphoria: * female volunteer without gender dysphoria according to DSM-V criteria (axis I), confirmed by MINI evaluation
  * volunteer aged 18 to 60 years
  * volunteer with normal or corrected vision
  * volunteer without mental defect
  * volunteer without neurological impairment
  Interventions: Other: Psychiatric evaluations

INTERVENTIONS:
Other: Psychiatric evaluations — At different time points, several psychiatric evaluations will be performed on patients and volunteers for study purposes
  Other Names: Electroencephalography; Double Mirror Test; Mini International Neuropsychiatric Interview; Montgomery-Åsberg Depression Rating Scale; Hamilton Rating Scale for Depression

SUMMARY:
Gender dysphoria is manifested by an internal tension between biological sex and gender, that is, by a non-congruence, in the subjects who suffer from it, between their sex of birth and their social gender identity.

DETAILED DESCRIPTION:
Gender dysphoria is manifested by an internal tension between biological sex and gender, that is, by a non-congruence, in the subjects who suffer from it, between their sex of birth and their social gender identity. Gender dysphoria is accompanied by the often overwhelming need for a hormonal or even hormone-surgical transition. Gender dysphoria is very often characterized by fluctuating mood sadness, irritability, obsessionality. An improvement in the quality of life after medical treatment (hormone therapy) and gender reassignment surgery has been described in the literature. Morphological similarities have been found between the brains of women and the brains of so-called transgender women, as well as between the brains of transgender men and men. These morphological data are only very fragmentary and have not been supported by neuro-functional data. Self-awareness, which refers to the awareness that an individual has of his body, his image and his own identity, is partly underpinned, at the brain level, by the activation of the Default Mode Network (DMN) at rest, in non-pathological conditions. The conflict between the internal perception of the own body and its objective representation could result in a change in brain connectivity within the DMN, due in particular to changes in the activation of the temporo parietal junction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gender dysphoria
* Without psychotropic
* Without hormono-therapy
* Without sexual surgery assignation

Exclusion Criteria:

* Any depression
* Any addiction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Contact sponsor for more details
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-03-26 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Contribution of temporal parameters of microstates C, D, E and F | Week 1 to Week 24
  The proportion of the total time spent in microstates of class C,D,E and F
Duration of temporal parameters of microstates C, D, E and F | Week 1 to Week 24
Mean-Global Field Power temporal parameters of microstates C, D, E and F | Week 1 to Week 24
Occurrence of temporal parameters of microstates C, D, E and F | Week 1 to Week 24
Cortical voxel activity from source reconstruction analysis, using electroencephalogram during Double Mirror Test (D.M.T). | Week 1 to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided